CLINICAL TRIAL: NCT06511973
Title: A 21-Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of BAY H006689, Naproxen 10% Topical Gel in Healthy Subjects Using a Cumulative Irritant Patch Test Design
Brief Title: A Study to Learn About Whether BAYH006689 Causes Skin Irritation When Applied as a Topical Gel in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 22641
Record Dates: First submitted 2024-07-11; First posted 2024-07-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain; Healthy Volunteers
MeSH Terms: conditions — Pain | interventions — Naproxen; Sodium Chloride; long-chain-aldehyde dehydrogenase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The treatments (IPs and control) will not be blinded to investigative personnel involved in the preparation/application and removal of treatments. However, the Investigator and trained evaluator involved in the evaluation of responses, will remain blinded during the course of the study until Database Lock and finalization of the Statistical Analysis Plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAYHO06689 (Experimental): Topical application of BAYH006689 naproxen 10% topical gel on the intact skin
  Interventions: Drug: Naproxen (BAYH006689)
- Placebo (Placebo Comparator): Topical application of placebo gel which contains 0% of naproxen on the intact skin
  Interventions: Drug: Placebo Gel
- Negative control (Placebo Comparator): Topical application of the sterile 0.9% saline (negative control) on the intact skin
  Interventions: Drug: A solution of 0.9% Saline
- Positive control (Active Comparator): Topical application of the 0.2% sodium lauryl sulfate (SLS) (positive control) on the intact skin
  Interventions: Drug: A solution of 0.2% SLS

INTERVENTIONS:
Drug: Naproxen (BAYH006689) — BAYH006689 gel will be dispensed directly on the patch
  Arms: BAYHO06689
Drug: Placebo Gel — Placebo gel will be dispensed directly on the patch
  Arms: Placebo
Drug: A solution of 0.9% Saline — 0.9% Saline will be dispensed directly on the patch
  Arms: Negative control
Drug: A solution of 0.2% SLS — 0.2% SLS will be dispensed directly on the patch.
  Arms: Positive control

SUMMARY:
Researchers are looking for a better way to treat muscle and joint pains. Researchers have seen that medicines which help reduce pain and inflammation could be safer when applied directly to the skin, called topical application, than when taken by mouth. However, recent studies have found that using these medications on the skin can sometimes cause skin reactions such as redness, itching, or irritation in the area where the medication is applied.

BAYH006689 topical gel is under development for the treatment of muscle and joint pains.

In this study, participants will be healthy and will not benefit from BAYH006689. However, the study will provide information about how to test BAYH006689 in future studies with people who have muscle and joint pain.

The main purpose of this study is to check whether BAYH006689 topical gel causes any irritation to the skin in healthy participants using a patch test called cumulative irritant patch test design. To do this, researchers will apply gel to participants' skin once a day for 21 days. Skin reactions will be assessed using a scale which will provide a score for redness, swelling, and other signs of skin irritation.

In this study, researchers will randomly assign 4 sites adjacent to each other, on the back of the participants' bodies just below the shoulder blades.

The following treatment gels will be applied using a patch.

* BAYH006689
* Placebo, which looks like the study drug, but does not have any medicine in it.
* 0.2% sodium lauryl sulfate (is a common ingredient in personal care products and when in contact with skin it could cause some skin irritation)
* 0.9% saline

Each participant will be in this study for 22 days, which includes:

* a visit to the clinic within 21 days of the study start, to confirm if the participant can take part in the study.
* participants will receive their assigned treatment gels at the identified skin site for 21 days.
* an end of study visit on Day 22, during which the researchers will remove the designed patches and assess any signs of skin irritation.

During the study, the doctors and their study team will:

* do physical examinations
* check participants' health by performing urine tests
* ask the participants questions about how they are feeling and what adverse events they are having An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Is 18 years of age or older
* Free of any systemic or dermatological disorder that may interfere with results or increase risk of adverse events (AEs)

Exclusion Criteria:

* Has a condition and/or is using medications that may interfere with the study results
* Pregnant or planning to get pregnant or breastfeeding
* Is currently participating in any clinical testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Skin sensitization potential measured by the mean and total cumulative irritancy score | 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.